CLINICAL TRIAL: NCT00851747
Title: A Randomized, Double-Blinded, Study of the Efficacy of Subcutaneous Phosphatidylcholine and Deoxycholate Injections for Localized Fat Removal
Brief Title: A Study of the Efficacy of Subcutaneous Phosphatidylcholine and Deoxycholate Injections for Localized Fat Removal
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CCF2
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blind

ARMS (3):
- C Phosphatidylcholine Deoxycholate (Experimental): Phosphatidylcholine Deoxycholate Injections. Group C will receive only study drug injections
  Interventions: Drug: Phosphatidylcholine Deoxycholate
- A Saline (Placebo Comparator): Group A will serve as a control and will receive only injections of saline as a placebo.
  Interventions: Drug: Saline
- B PhosphatidylcholineDeoxycholate/Saline (Active Comparator): Group B will receive saline injections on one side of the body and receive study drug injections on the contralateral side.
  Interventions: Drug: Phosphatidylcholine Deoxycholate; Drug: Saline

INTERVENTIONS:
Drug: Phosphatidylcholine Deoxycholate — Group A will serve as a control and will receive only injections of saline as a placebo. Group B will receive saline injections on one side of the body and receive study drug injections on the contralateral side. Group C will receive only study drug injections
  Other Names: Lipodissolve; Lipolight
  Arms: B PhosphatidylcholineDeoxycholate/Saline; C Phosphatidylcholine Deoxycholate
Drug: Saline — Group A will serve as a control and will receive only injections of saline as a placebo. Group B will receive saline injections on one side of the body and receive study drug injections on the contralateral side. Group C will receive only study drug injections
  Other Names: salt solution
  Arms: A Saline; B PhosphatidylcholineDeoxycholate/Saline

SUMMARY:
The primary objective of this study is to determine the efficacy of phosphatidylcholine and deoxycholate subcutaneous injections for localized fat removal.

Subcutaneous injections of the study drug will be efficacious in decreasing localized fat deposits due to the known fat necrosis effects on fat tissue after study drug tissue incubation.

DETAILED DESCRIPTION:
This study is a randomized, double-blind study of 21 subjects. Participants in this study will be healthy, non-obese (BMI <30) subjects over 25 with two localized, symmetrical, and contralateral areas of fat deposition on the abdomen or flanks and on the buttocks or thighs that have proven resistant to diet and exercise. Each participant will be randomized to one of three groups and will receive 4 series of injections two weeks apart. Multiple injections will be placed in the subdermal fat layer from 1-1.5 cm apart depending on the size of the treatment area.

Group A will serve as a control and will receive only injections of saline as a placebo. Group B will receive saline injections on one side of the body and receive study drug injections on the contralateral side. Group C will receive only study drug injections. The study sites will include a symmetric, contralateral area of localized fat deposit on both the upper and lower torso. Clinical evaluations will be performed at each visit. Hematologic and ultrasonographic evaluations will be performed at baseline, at the 3rd treatment (Week 4), and at 6 month follow-up. Histologic evaluations will be performed on select individuals at baseline and at the 3rd treatment (Week 4) visit.

ELIGIBILITY:
Inclusion Criteria:

* Age 25 and over
* BMI of 18.5-29.99
* Two localized areas of fat deposition on the upper and lower torso that have failed on self-reported diet and exercise
* The subject is in good health
* The subject has the willingness and the ability to understand and provide informed consent

Exclusion Criteria:

* Under 25 years of age
* Pregnancy or Lactation
* BMI≥ 30
* Subjects with known eating disorders or a history of weight loss/gain of 5 pounds or more within the past 6 months
* Subjects with hepatrophy, nephopathy, diabetes, hyperthyroidism, neoplasias, AIDS or other immuno-compromised illness, allergies to eggs or soy, poorly controlled hypertension, or autoimmune disease
* Subjects currently taking blood thinners or who have had chemotherapy or radiation within the last 6 months
* Subjects with an open, non-healing sore or infection near site of injection
* Subjects with active eczema or psoriasis
* Subjects who are unable to understand the protocol or to give informed consent
* Subjects with mental illness

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-02; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- B PhosphatidylcholineDeoxycholate/Saliine: Group B will receive saline injections on one side of the body and receive study drug injections on the contralateral side
- C Phosphatidylcholine Deoxycholate: Phosphatidylcholine Deoxycholate Injections
  Group C will receive only study drug injections
Period: Overall Study
Arm/Group | A Saline | B PhosphatidylcholineDeoxycholate/Saliine | C Phosphatidylcholine Deoxycholate
Started | 6 | 6 | 6
Completed | 0 | 0 | 0
Not Completed | 6 | 6 | 6
Not completed — Physician Decision | 6 | 6 | 6

BASELINE CHARACTERISTICS:
Population: No analysis completed. PI left the institution
Groups:
- C Phosphatidylcholine Deoxycholate: Phosphatidylcholine Deoxycholate Injections
- B PhosphatidylcholineDeoxycholate/Saline: Group B will receive saline injections on one side of the body and receive PhosphatidylcholineDeoxycholate injections on the contralateral side.
- Total: Total of all reporting groups
Arm/Group | C Phosphatidylcholine Deoxycholate | A Saline | B PhosphatidylcholineDeoxycholate/Saline | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Categorical [Count of Participants; unit: Participants] — Population: PI left institution no data available.
Sex: Female, Male [Count of Participants; unit: Participants] — Population: No analysis completed. PI left the Institution

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Phosphatidylcholine and Deoxycholate Subcutaneous Injections for Localized Fat Removal.
Description: The primary objective of this study is to determine the efficacy of phosphatidylcholine and deoxycholate subcutaneous injections for localized fat removal. Subcutaneous injections of the study drug will be efficacious in decreasing localized fat deposits
Time Frame: 1 year
Population: PI left institution and no data is available.
Groups:
- Subcutaneous Injections: Phosphatidylcholine Deoxycholate Injections
  Phosphatidylcholine Deoxycholate: Group A will serve as a control and will receive only injections of saline as a placebo. Group B will receive saline injections on one side of the body and receive study drug injections on the contralateral side. Group C will receive only study drug injections
  Saline: Group A will serve as a control and will receive only injections of saline as a placebo. Group B will receive saline injections on one side of the body and receive study drug injections on the contralateral side. Group C will receive only study drug injections
Arm/Group | Subcutaneous Injections | Saline
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- C Phosphatidylcholine Deoxycholate: Group C will receive only Phosphatidylcholine Deoxycholate injections
Arm/Group | C Phosphatidylcholine Deoxycholate | A Saline | B PhosphatidylcholineDeoxycholate/Saline
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6

LIMITATIONS AND CAVEATS:
PI left institution, no data available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes